CLINICAL TRIAL: NCT02563041
Title: Comparative Effectiveness of 30% Trisodium Citrate and Heparin Lock Solutions in Preventing Infection and Dysfunction of Hemodialysis Catheters: a Randomized Controlled Trial (CITRIM Trial)
Brief Title: Comparative Effectiveness of 30%TSC and Heparin Lock Solution in Hemodialysis Catheters
Acronym: CITRIM
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Catholic University of Pelotas (Other)
Responsible Party: Principal Investigator, Maristela Bohlke, MD PhD, Catholic University of Pelotas
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: UCPel
Record Dates: First submitted 2015-09-23; First posted 2015-09-29 (Estimated); Last update posted 2015-09-29 (Estimated); Status verified 2015-09

CONDITIONS: Catheter Related Infection
MeSH Terms: conditions — Catheter-Related Infections | interventions — trans-sodium crocetinate; trisodium citrate; Heparin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 30%TSC (Experimental): After each hemodialysis (HD) session, the catheter lumens were flushed with 0.9% sodium chloride and locked with a volume of 30%TSC solution exactly equivalent to the catheter internal lumen.
  Interventions: Drug: 30% TSC
- Heparin 5000 U/mL (Active Comparator): After each hemodialysis (HD) session, the catheter lumens were flushed with 0.9% sodium chloride and locked with a volume of unfractionated sodium heparin 5000 U/mL solution exactly equivalent to the catheter internal lumen.
  Interventions: Drug: Heparin

INTERVENTIONS:
Drug: 30% TSC — The patients were randomly assigned to have their catheter locked with either unfractionated sodium heparin 5000 U/mL or 30% trisodium citrate.
  Other Names: 30% trisodium citrate
  Arms: 30%TSC
Drug: Heparin — The patients were randomly assigned to have their catheter locked with either unfractionated sodium heparin 5000 U/mL or 30% trisodium citrate.
  Other Names: unfractionated sodium heparin 5000 U/mL
  Arms: Heparin 5000 U/mL

SUMMARY:
BACKGROUND: Central venous catheters (CVC) are the only option when hemodialysis is needed for patients without definitive vascular access. However, CVC use is associated with complications such as infection, thrombosis, and dysfunction, leading to higher mortality and expenditures. The aim of this study was to compare the effectiveness of 30% trisodium citrate (TSC30%) with heparin as CVC lock solution in preventing catheter-related bloodstream infections (CRBSI) and dysfunction in hemodialysis patients. METHODS: Randomized, double-blind controlled trial comparing the event-free survival of non-tunneled CVC locked with heparin or TSC30% in adult hemodialysis patients.

DETAILED DESCRIPTION:
METHODS Study Design This double blind randomized controlled trial (RCT) was conducted from July 2012 until July 2014 in the dialysis and transplantation unit of a Brazilian university hospital. The patients were randomly assigned to have their catheter locked with either unfractionated sodium heparin 5000 U/mL or 30% trisodium citrate. The randomization was performed through a computer-generated list of random numbers in blocks of six. Patients and investigators were unaware of the treatment assignments. Allocation concealment was performed using opaque, sealed envelopes for assignment.

After each hemodialysis (HD) session, patients assigned to 30%TSC had their catheter lumens flushed with 0.9% sodium chloride and locked with a volume of 30% TSC solution equivalent to the catheter internal lumen. Patients assigned to heparin had their catheter lumens flushed with 0.9% sodium chloride and locked with a volume of 5000 U/mL heparin equivalent to CVC internal lumen. Catheter care was according to international guidelines, including strict asepsis on insertion and exit-site dressing changes after each HD session by staff wearing masks and sterile gloves.

SELECTION OF PATIENTS Patients were eligible for enrollment in the RCT when they were older than 18 years and had chronic or acute renal failure that required hemodialysis through a catheter. Patients admitted to the intensive care ward, receiving a tunneled catheter, with suspected heparin-induced thrombocytopenia, allergy to heparin or TSC30%, with systemic or localized infection or pregnant women were excluded. The site of insertion and specific type of catheter were decided by the interventionist physician.

MAIN OUTCOMES Catheter related bloodstream infection (CRBSI): CRBSI was defined as fever and/or chills during a dialysis session and at least one positive blood culture, with no other obvious cause of infection after careful clinical examination. The management of the CRBSI was performed according to guidelines. Empirical antibiotic therapy was immediately given. The catheter was removed if there was isolation of S. aureus or fungus, or there was no clinical recovery within 48 hours of antibiotic treatment.

Catheter dysfunction: Dysfunction was defined as a persistent inability to obtain a blood flow above 200 mL/min. In this situation, the catheter was removed or exchanged over guidewire.

OTHER PREDICTORS Patients-related: Data was also collected about age, gender, skin color, presence of diabetes, diagnosis of CKD or acute kidney injury, and hemodialysis vintage.

Catheter-related: Site of insertion (jugular, subclavian or femoral vein), and ordinal number of catheter in the same patient (considering only the study period).

STATISTICAL ANALYSIS Calculation of the required sample size was based on main outcomes. It was assumed that the group with heparin lock would have a rate of catheter-related bloodstream infection of 150% greater than that of catheters with TCS30% lock. With a two-sided test, and an alfa error of 5% and 80% of power, it was required 112 catheters for each group.

The primary analysis was made through survival analysis with Cox proportional hazard regression. Initially the investigators proceed to univariate analysis using Kaplan-Meier curves and log rank test for the categorical variables, and univariate Cox regression for continuous variables. The predictors which have a p-value lower than 0.25 in univariate analysis were included in final model. Interactions were checked for any possible association of predictors. The likelihood ratio test was used for compare nested with full models. The proportionality of predictors was verified by introduction of time-dependent variables in the model. If any predictor violates the proportionality assumption, the analysis would be stratified for that predictor. Well-functioning catheters at the end of the study period, catheters removed because patients acquired functional arteriovenous fistula, renal function recovery, changed to peritoneal dialysis or had transplantation were analyzed as censored data. The analysis was all done on intention-to-treat base. All reported p-value are two sided. The analysis was performed using the STATA 11.2 statistical software (Stata Corporation, College Station, TX, USA)

ETHICAL ASPECTS The study protocol was approved by the local review board. Written informed consent was obtained from all patients before enrollment.

ELIGIBILITY:
Inclusion Criteria:

* patients older than 18 years and
* with chronic or acute renal failure and
* requiring hemodialysis through a catheter.

Exclusion Criteria:

* patients admitted to the intensive care ward,
* receiving a tunneled catheter,
* patients with suspected heparin-induced thrombocytopenia,
* patients with allergy to heparin or TSC30%,
* patients with systemic or localized infection
* pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 179 (Actual)
Dates: Start 2012-07; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Catheter related bloodstream infection | through study completion, an average of 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Maristela Bohlke, MD, PhD, Principal Investigator — Catholic University of Pelotas

REFERENCES:
- [Derived] Correa Barcellos F, Pereira Nunes B, Jorge Valle L, Lopes T, Orlando B, Scherer C, Nunes M, Araujo Duarte G, Bohlke M. Comparative effectiveness of 30 % trisodium citrate and heparin lock solution in preventing infection and dysfunction of hemodialysis catheters: a randomized controlled trial (CITRIM trial). Infection. 2017 Apr;45(2):139-145. doi: 10.1007/s15010-016-0929-4. Epub 2016 Aug 29. PMID 27573387